CLINICAL TRIAL: NCT05959330
Title: Effects of Neural Tension Versus Neural Sliding Technique on Pain, Cervical Muscle Endurance and Hand Grip Strength in Unilateral Cervical Radiculopathy
Brief Title: Effects of Neural Tension Versus Neural Sliding Technique on Cervical Radiculopathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RiphahIU Sehar Fatima
Record Dates: First submitted 2023-03-31; First posted 2023-07-25 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Cervical Radiculopathy
Keywords: Slider; Tensioner Neurodynamic Mobilization; Cervical Radiculopathy; Hand Grip Strength; Numeric Pain Rating Scale
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neural Tension Technique(ulnar, median, radial) (Experimental): Neural Tension Technique for 4 weeks (6 successive sessions). Three sets will be provided in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment
  Interventions: Other: Neural Tension Technique(ulnar, median, radial)
- Neural Slider Technique (ulnar, median, radial) (Experimental): Neural Slider Technique for 4 weeks (6 successive sessions). Three sets will be provided in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment
  Interventions: Other: Neural Slider Technique (ulnar, median, radial)
- Neural Tension Technique and Neural Sliding Technique(ulnar, median, radial) (Experimental): Neural Tension and Sliding Technique for 4 weeks (6 successive sessions). Three sets will be provided in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment
  Interventions: Other: Neural Tension Technique and Neural Sliding Technique(ulnar, median, radial)

INTERVENTIONS:
Other: Neural Tension Technique(ulnar, median, radial) — Neural Tension Technique for 4 weeks (6 successive sessions). Three sets will be provided in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment
  Arms: Neural Tension Technique(ulnar, median, radial)
Other: Neural Slider Technique (ulnar, median, radial) — Neural Slider Technique for 4 weeks (6 successive sessions). Three sets will be provided in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment
  Arms: Neural Slider Technique (ulnar, median, radial)
Other: Neural Tension Technique and Neural Sliding Technique(ulnar, median, radial) — Neural Tension and Sliding Technique for 4 weeks (6 successive sessions). Three sets will be provided in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment
  Arms: Neural Tension Technique and Neural Sliding Technique(ulnar, median, radial)

SUMMARY:
The aim of this research is to find the effects of neural tension versus neural sliding technique on pain, cervical muscle endurance and hand grip strength in unilateral cervical radiculopathy. It will be a randomized controlled trial in which participants selected through non probability convenience sampling with age from 18 to 65 years having unilateral cervical radicular pain in upper limb since 3 months and any two of the following positive test Spurling's test, Distraction test and Upper Limb Tension Test. Participants will be randomly allocated, into three groups (A, B, and C). On the contrary, patients with any orthopedic or neurological conditions of cervical spine and shoulder joint, malignancy, cervical surgeries and bilateral cervical radiculopathies will be excluded from the study. Baseline measurement of all groups will be taken by using Numerical Pain Rating Scale (NPRS) for pain, Cranio-cervical Flexion Test for endurance and Hand-Held Dynamometer for hand grip strength. Group A will receive 7 neural tension technique, Group B will receive neural sliding technique, while Group C will receive both neural tension technique and neural sliding technique for 4 weeks (6 successive sessions). Both techniques (slider and tensioner) will be provided three sets in every session; Each set will be performed in a slow, oscillatory manner with 10 seconds rest between the sets. Posttest measurement will be taken after 4 weeks of treatment. SPSS 21 software will be used for data entry and analysis.

DETAILED DESCRIPTION:
Cervical radiculopathy also known as "pinched nerve", is a neurological condition caused by compression of the cervical spine nerve and roots. It is basically a lower motor neuron and sensory demonstration of neurological dysfunction of the involved cervical nerve root. Cervical radiculopathy is most commonly caused by the herniation of the cervical spine intervertebral disc or any space-occupying lesion that may lead to nerve root inflammation or impingement. Other common causes of cervical radiculopathy are spondylosis, trauma, osteoporosis, cervical instability, and sometimes oncological issues. Such problems either directly compress the cervical nerve roots or narrow the space of the vertebral foramen from where the cervical nerve root emerges which leads to neuritis, hypoxia, ischemia, fibrosis, edema, or decreased nerve mobility. Cervical radiculopathy has an average annual incident rate of 83 per 100,000 of the population with an increased prevalence in the fourth and fifth decade of life.

According to studies, the most commonly affected cervical nerve root is C7 followed by the C6 and C8. The clinical manifestation of cervical radiculopathy is quite broad involving motor and sensory changes in the upper extremity. Patients with cervical radiculopathy usually experience loss of sensation, tingling, numbness, motor defects in the neck and sometimes in the scapula, and pain in the arm and hand along the pathway of the nerve depending upon the location of the affected nerve root. The pain can be radiated both bilaterally and unilaterally into the arms, however, the prevalence of bilateral cervical radiculopathy is only 5 - 36%.

The symptoms of muscle weakness in the upper limb are often seen in patients with cervical radiculopathy. According to the principles of the kinetic chain, the upper limb is an integrated system consisting of different segments working together to accomplish the activities of daily living. In simpler words, the muscle weakness produced in any segment of the upper limb would result in generalized muscle weakness and ultimately decreased hand grip strength. To perform functional activities of daily living it is very important to maintain the grip strength of the upper extremity. But, to achieve the maximum grip strength the physical and physiological properties of nerve tissues need to be intact. Since reduced grip strength is often seen in patients with cervical radiculopathy, it becomes essential to administer an appropriate technique to rehabilitate its strength

Manual therapy techniques are considered effective in the treatment of cervical radiculopathy. Neurodynamic mobilization has been considered effective as a conservative management approach for the treatment of upper quadrant pain. It restores homeostasis in and around the neural tissues by improving the mechanical and neurophysiological integrity of the peripheral nerves, thus reducing pain and disability. Slider and tensioner are the two most commonly used neural mobilization techniques and a biomechanical distinction can be made between these two techniques. Neural mobilization plays an important role in returning to normal functional activities by restoring the range of motion and extensibility of the nervous system

Neurodynamic mobilization restores the neural tissues' ability to resist tension and stress by promoting the restoration of normal physiological function, decreasing pain, and improving function. The slider neurodynamic mobilization causes sliding movement in the neural tissue in correspondence to the nearby structures; distributing the compression and tension along the entire nervous instead of one particular region. On the other hand, tensioner neurodynamic mobilization causes tension in the neural tissue without surpassing the tissue elastic capacity that enhances nerve's viscoelastic properties. This procedure is done by taking the nerve, in the end, range of movement (elongated position), maintaining the position for a short duration, and then fully releasing the tension.

A systematic review of a randomized control trial was done by Papacharalambous C et al. in 2022 to evaluate the effectiveness of slider and tensioner neural mobilization techniques in the management of upper quadrant pain. The results of the study concluded that slider and tensioner neural mobilization techniques are quite effective in reducing pain in certain musculoskeletal conditions. Moreover, the results revealed that slider neural mobilization technique is more effective in the treatment of acute conditions than tensioner neural mobilization.

A randomized clinical trial was conducted by Shou MK et al. in 2022, to determine the effects of neural slider and contralateral cervical lateral glide in athletes with cervicobrachial pain syndrome. Thirty patients were recruited in the study that were divided into groups. One group received neural slider technique whereas the other received contralateral cervical lateral glide. The results revealed that both techniques are effective in improving pain and functional disability. However, the contralateral cervical lateral glide is more effective than the neural mobilization technique for patients with cervicobrachial pain syndrome.

Raval MM et al. conducted a comparative study in 2022 to determine the effect of neural sliding technique versus neural sliding technique on functional disability and pain in patients with cervical radiculopathy. A total of thirty patients were recruited for the study and later divided into two equal groups. Group A received neural tension mobilization while Group B received neural sliding mobilization. Outcome measure tools Numeric Pain Rating Scale, Neck Disability Index, and Patient Specific Functional Scale were used to access the patient before and after the treatment. The results of the study concluded that tensioner neurodynamic mobilization is more effective in reducing functional disability and pain than slider neurodynamic mobilization.

ELIGIBILITY:
Inclusion Criteria:

* • Unilateral radicular pain in upper limb since 3 months(10)

  * Any two of the following tests positive: Spurling's test, Distraction test, Upper Limb Tension Test

Exclusion Criteria:

* • Any orthopedic or neurological conditions of cervical spine and shoulder joint

  * Hypermobility of cervical spine
  * Malignancy
  * Vertebro-basilar insufficiency
  * Patients undergone cervical surgeries
  * Patients with bilateral cervical radiculopathies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | Changes from baseline Numeric Pain Rating Scale (NPRS) at 1 months
  Numeric Pain Rating Scale is a subjective outcome measure tool that is used to measure intensity of pain in adults. It is a numeric version of Visual Analogue Scale. NPRS is a unidirectional 11- point scale that ranges from 0 to 10. With "0" indicating the 'no pain at all' and "10" indicating the 'the worst pain imaginable'. The NPRS can be administered either graphically or verbally. The respondent is asked to indicate the numeric value that describes their current pain intensity best
Hand-Held Dynamometer | Changes from baseline Hand-Held Dynamometer (HHD) at 1 months
  The patient will be asked to sit on a straight back chair with his/her feet flat on the floor. The affected shoulder was to be maintained at 0º of flexion, abduction and rotation, elbow flexed to 90º, forearm rested in a neutral position with the wrist in minimal extension and ulnar deviation.
  On achieving the standardized arm position, the dynamometer set at the second handle space was given to subjects who were then advised to perform 3 maximum gripping efforts for 5 seconds. A 15 second rest period was given to prevent fatigue effects.
  While performing each trial, each patient was instructed by the assessor as follows: "Squeeze the handle as hard as possible". The mean value of the 3 efforts (measured in pounds) was evaluated for the analysis of grip strength. The patients were not allowed to see their score in each trial. No visual and verbal encouragement was given for achieving the maxi-mum capable grip strength
Cervico-cranial Flexion Test (Blood Pressure Cuff) | Changes from baseline Cervico-cranial Flexion Test (CCFT) at 1 months
  A blood pressure cuff is inflated to 20 mmHg and is placed between the lordotic curve and the surface of the table. While keeping the back of the head stable, the patient performs cranial cervical flexion in a graded fashion in 5 increments (22, 24, 26, 28, and 30 mmHg). Each position is held for 10 seconds with 10 seconds rest between increments. The cranial cervical flexion is performed by a head nod in the upper cervical spine. Make sure the patient's jaw is relaxed, so that there is no platysma, hyoid muscle, or sternocleidomastoid recruitment.
  The test is ended when the pressure decreases >20% or when substitution occurs during the head nod. Normal response is achieving 26-30 mmHg.[

CONTACTS AND LOCATIONS:
Overall Officials: Sehar Fatima, DPT, Principal Investigator — Riphah International University
Locations (1):
- Service Hospital Lahore, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang KC, Lee HS, Lee JH. Cervical Radiculopathy Focus on Characteristics and Differential Diagnosis. Asian Spine J. 2020 Dec;14(6):921-930. doi: 10.31616/asj.2020.0647. Epub 2020 Dec 22. PMID 33373515